CLINICAL TRIAL: NCT06387836
Title: Impact of Desflurane Versus Isoflurane on Early Cognitive Function of the Elderly Undergoing Lumbar Surgery: A Randomized Clinical Trial
Brief Title: LINC01844 as a Diagnostic Biomarker for POCD in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2024-063
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: postoperative cognitive dysfunction; long intergenic non-coding RNA; prediction biomarker
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iso anesthesia (Active Comparator): Patients in this group are under anesthesia with isoflurane.
  Interventions: Drug: Isoflurane 0.8 MAC
- Des anesthesia (Active Comparator): Patients in this group are under anesthesia with desflurane.
  Interventions: Drug: Desflurane 0.8MAC

INTERVENTIONS:
Drug: Isoflurane 0.8 MAC — Patients in this group will be anesthetized using isoflurane with the depth of 0.8~1.0MAC during the operation.
  Arms: Iso anesthesia
Drug: Desflurane 0.8MAC — Patients in this group will be anesthetized using desflurane with the depth of 0.8~1.0MAC during the operation.
  Arms: Des anesthesia

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a common complication after surgery that is associated with more adverse events and death. The goal of this randomized, controlled clinical study is to learn about the impact of different inhalation anesthetics may have on the elderly in terms of POCD and diagnosis performance of long intergenic non-coding RNA(LINC01844) level in blood of older people for POCD. The main question it aims to answer is: Dose the desflurane have less influence on the elderly's cognitive function in comparison with isoflurane？Does the relative level of LINC01844 in blood help diagnose POCD of older people after surgery? Participants undergoing elective lumbar decompression and fusion will finish neuropsychological evaluations one day before and 1st, 3rd and 5th day after surgery. At the same timepoint, the relative level of LINC01844 in blood will also be tested.

DETAILED DESCRIPTION:
Trial design This single-center, randomized, controlled trial will enroll patients undergoing elective lumbar decompression and fusion at Zhongshan Hospital Fudan University, Shanghai, China. Written informed consent is obtained from all the participants. By Feb 21, 2024, the trial was approved for Zhongshan Hospital, Fudan University (China) with the approval number B2024-063R.

Anesthesia After the patients entered the operating room, the vital signs are monitored, the patients are given oxygen inhalation (> 8L/min). General anesthesia is induced with sufentanil (0.2ug/kg), propofol [target controlled infusion (TCI) at plasma concentration of 3ug/ml) , remifentanil(TCI at plasma concentration of 3 ng/ml) and rocuronium (0.6mg/kg). The narcotic and vasoactive drugs are used during the operation according to anesthesia depth, the blood pressure, and respiratory parameters. A patient-controlled intravenous analgesia (PCIA) pump (sufentanil 250ug, and ramosetron 0.6mg) is connected after the surgery.

Detection and preparation of LINC01844 Total RNA is extracted from peripheral blood samples using TRIzol LS (Invitrogen, USA) according to the instructions from the manufacturer. Briefly, after homogenizing the blood sample (250 μL) with TRIzol LS regent (750 μL), chloroform (200 μL) is added for further analysis. The sample is centrifuged at 12,000 × g, 4˚C for 15 min, then the aqueous phase containing the RNA is transferred to a new tube and isopropanol (0.5 mL) is added for RNA precipitation. The RNA pellet is washed by 75% ethanol (1 mL), and finally resuspended in RNase free water (10-20 μL), the RNA quality is determined with NanoDrop2000. An optical density ratio of 260/280 >1.80 is an indication that the sample could be used in subsequent experiments. Next, we use M-MLV reverse transcriptase (Promega, USA) for the synthesis of cDNA. A real-time quantitative polymerase chain reaction (qRT-PCR) was utilized for the final analysis according to the instructions from the SYBR Green PCR Master Mix Kit (Qiagen). The PCR parameters: 95˚C for 10 min; 45 cycles at 95˚C for 15 s, 60˚C for 30s, and 72˚C 30s. GAPDH is chosen as a reference gene, fold change (2 -44Ct ) is utilized to analyze LINC01844 relative levels.

Neuropsychological test evaluation and POCD assessment One day before surgery, patients will be assessed for depression using the patient health Questionnaire-9 (PHQ-9), while patients with previous severe cognitive impairment are excluded using the mini mental state examination (MMSE) (MMSE score < 24). A battery of neuropsychological tests will be performed 1 day before operation and 1st, 3rd and 5th day after operation to evaluate the cognitive function of patients, including Hopkins auditory learning test-revised (HALT-R), brief visuospatial memory test-revised (BVMT-R), trail making test (TMT), digit span test (DST), digital symbol substitution test (DSST) and verb and graph recall test. All these tests are performed in a quiet environment by a trained doctor who is blinded to the surgical procedure and blood sample. At the same time, 20 healthy volunteers without surgery will be recruited as the control group, with age, sex and education years matched. The neuropsychological test will be performed in control group to determine the normal reference value of cognitive function, with the same interval. Baseline scores and learning outcomes were subtracted from each neuropsychological test score according to the international guidelines for the study of postoperative cognitive impairment, and divided by the standard deviation of baseline scores in the control group. The result was designated a Z score. When at least two Z scales are greater than 1.961, POCD was considered.

Study visits and data collection Patients will be visited preoperatively and postoperative day (POD) 1 and 3 and 5. The patients will be screened according to the inclusion criteria. All patients meeting the inclusion criteria will be registered in a screening log file. The investigators will explain the course and purpose of the study and provide written information on the study. Patients willing to participate in the study will be required to provide written informed consent.

Data will be registered in both the paper case report form (CRF) and the electronic case report form (eCRF) on electronic data capture (EDC) system by trial or clinical personnel under the supervision of the trial site investigators. In the case of inconsistency, the paper CRF will be used as a gold standard.

Handling of data Two members of the research team will perform study monitoring. Remote monitoring will be performed to signal early aberrant patterns, issues with consistency, credibility, and other anomalies. Patient data will be collected in pseudonymous form using a patient (identification) number composed of four three digits. Study data will be collected and managed using an investigator-initiated trial EDC (IIT-EDC) tools. IIT-EDC is a password-protected, intranet-based application designed to support data record for research studies (website: http://10.15.7.137). Full access to the final trial dataset will be granted to selected investigators. All original records, including consent forms, reports of suspected unexpected serious adverse events (SAE), and relevant correspondences, will be archived at the trial sites for 10 years. The clean trial database file will be anonymized and maintained for 10 years.

Safety All adverse events (AE) thought to be related to the trial will be reported to the trial coordinating center. According to local laws and regulations, the participants may receive free treatment provided by our unit or be compensated if any injury related to this study does occur, and all suspected unexpected SAEs will be reported to the data monitoring and safety committee (DMSC). The DMSC is independent of the trial investigators and will perform an ongoing review of safety parameters and overall study conduct. The DMSC comprises two independent experts in large-scale clinical trials and one independent statistician. The DMSC will be responsible for safeguarding the interests of the trial participants, assessing the safety and efficacy of the interventions during the trial, and monitoring the overall conduct of the clinical trial. To enhance the integrity of the trial, the DMSC may also formulate recommendations relating to the recruitment/retention of participants, their management, improving adherence to protocol-specified regimens and retention of participants, and procedures for data management and quality control.

Statistical analysis Sample size -To verify the different influence on postoperative cognitive function for older people after surgery between isoflurane and desflurane, a test for two-proportions model is used to calculate the sample size. Based on results from preliminary trial, the incidence of POCD was 15% and 40% for desflurane group and isoflurane group, respectively. Sample size was calculated by PASS (version 11.0). For power of 80% and level of significance of 5% against the one-sided alternative hypothesis, 38 participants are required for one group. Expecting 10% drop-out of participants, a sample size of total 86 is required.

Analysis - Kolmogorov-Smirnov test will be used to assess the normal distribution of continuous data. The baseline characteristics will be expressed as counts and percentages, means and standard deviations, or medians and interquartile ranges, as appropriate. The independent predictors of POCD were analyzed by binary logistic regression, and the results were expressed as odds ratios (ORs). The prediction performance of LINC01844 for POCD will be measured using ROC, and the results were determined by the 95% confidence intervals and AUC. No or minimal losses to follow-up for the primary and secondary outcomes are anticipated. The intention-to-treat (ITT, all randomly assigned cases) population is used for all outcomes analysis. The supportive analysis is based on full analysis set (FAS, all randomly assigned patients who receive lumbar decompression and fusion). Complete-case analysis will be performed for all outcomes. However, if more than 1% of missing data are found for the primary outcome, a sensitivity analysis using multiple imputations and estimating equation methods will be carried out.

Cleaning and locking of the database The datasets used and/or analyzed during the current study will be made available from the corresponding author upon reasonable request. The database will be locked immediately after all data are entered and all discrepant or missing data are resolved, or, alternatively, if all efforts have been employed and we consider that the remaining issues cannot be fixed. In this step, the data will be reviewed before database locking. The study database will then be locked and exported for statistical analysis. At this stage, permission for access to the database will be removed for all investigators, and the database will be archived.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to perform elective lumbar decompression and interbody fusion under general anesthesia;
* 65-85 years old;
* American Society of Anesthesiologists (ASA) physical status I-III level;
* Body mass index (BMI) between 20 Kg/m2 and 28 Kg/m2;
* From whom written informed consent is obtainable either from the patient or from a legal representative;

Exclusion Criteria:

* Patents with cognitive dysfunction preoperatively;
* Patents with verbal, visual and auditory defects;
* Patients with history of alcohol and/or drug abuse, or history of neurological and psychotic disorders;
* Patients with history of hospital admission and therapy within 30 days.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
incidence of POCD | From date of randomization until the date of telephone follow-up completed , assessed up to 2 months.
  The incidence of POCD is defined as the proportion of people who is diagnosed POCD at least once of the three times(on postoperative day 1, day 3 and day 5) in this group. POCD is diagnosed using the Z-score method. Patients were tested with a battery of 7 neurocognitive tests, and POCD was considered when the Z-score > 1.961in two or more tests .

SECONDARY OUTCOMES:
serum reactive protein-C | From date of randomization until the date of discharge , assessed up to 10 days.
  Serum reactive protein-C is measured by an ELISA kit
serum interleukin-6 | From date of randomization until the date of discharge , assessed up to 10 days.
  Serum interleukin-6 is measured by an ELISA kit
relative level of LINC01844 | From date of randomization until the date of discharge , assessed up to 10 days.
  Total RNA is extracted from blood samples using TRIzolLS (Invitrogen, USA) according to the manufacturer's instructions. The RNA concentration and purity were determined by NanoDrop2000, and the absorbance of 260/230>1.8 indicated that the RNA purity was higher. Then, reverse transcription (Promega, USA) and quantitative real-time polymerase chain reaction (qRT-PCR) were performed to analyze the expression of L INC01844.With GAPDH as the internal control, the fold change is expressed as 2-△△Ct.

CONTACTS AND LOCATIONS:
Overall Officials: Shengjin Ge, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There isn't an IPD plan yet. Full access to the final trial dataset will only be granted to selected investigators for publication issues.

REFERENCES:
- [Background] Pandin P, Estruc I, Van Hecke D, Truong HN, Marullo L, Hublet S, Van Obbergh L. Brain Aging and Anesthesia. J Cardiothorac Vasc Anesth. 2019 Aug;33 Suppl 1:S58-S66. doi: 10.1053/j.jvca.2019.03.042. PMID 31279354
- [Background] Cortese GP, Burger C. Neuroinflammatory challenges compromise neuronal function in the aging brain: Postoperative cognitive delirium and Alzheimer's disease. Behav Brain Res. 2017 Mar 30;322(Pt B):269-279. doi: 10.1016/j.bbr.2016.08.027. Epub 2016 Aug 17. PMID 27544872
- [Background] Mashour GA, Woodrum DT, Avidan MS. Neurological complications of surgery and anaesthesia. Br J Anaesth. 2015 Feb;114(2):194-203. doi: 10.1093/bja/aeu296. Epub 2014 Sep 8. PMID 25204699
- [Background] Iqbal F, Thompson AJ, Riaz S, Pehar M, Rice T, Syed NI. Anesthetics: from modes of action to unconsciousness and neurotoxicity. J Neurophysiol. 2019 Aug 1;122(2):760-787. doi: 10.1152/jn.00210.2019. Epub 2019 Jun 26. PMID 31242059
- [Background] Gitman M, Fettiplace MR, Weinberg GL, Neal JM, Barrington MJ. Local Anesthetic Systemic Toxicity: A Narrative Literature Review and Clinical Update on Prevention, Diagnosis, and Management. Plast Reconstr Surg. 2019 Sep;144(3):783-795. doi: 10.1097/PRS.0000000000005989. PMID 31461049
- [Background] Carr ZJ, Cios TJ, Potter KF, Swick JT. Does Dexmedetomidine Ameliorate Postoperative Cognitive Dysfunction? A Brief Review of the Recent Literature. Curr Neurol Neurosci Rep. 2018 Aug 6;18(10):64. doi: 10.1007/s11910-018-0873-z. PMID 30083844
- [Background] Zhang B, Tian M, Zhen Y, Yue Y, Sherman J, Zheng H, Li S, Tanzi RE, Marcantonio ER, Xie Z. The effects of isoflurane and desflurane on cognitive function in humans. Anesth Analg. 2012 Feb;114(2):410-5. doi: 10.1213/ANE.0b013e31823b2602. Epub 2011 Nov 10. PMID 22075020
- [Background] Schallner N, Ulbrich F, Engelstaedter H, Biermann J, Auwaerter V, Loop T, Goebel U. Isoflurane but not sevoflurane or desflurane aggravates injury to neurons in vitro and in vivo via p75NTR-NF-kB activation. Anesth Analg. 2014 Dec;119(6):1429-41. doi: 10.1213/ANE.0000000000000488. PMID 25329094
- [Background] Jiang J, Jiang H. Effect of the inhaled anesthetics isoflurane, sevoflurane and desflurane on the neuropathogenesis of Alzheimer's disease (review). Mol Med Rep. 2015 Jul;12(1):3-12. doi: 10.3892/mmr.2015.3424. Epub 2015 Mar 4. PMID 25738734
- [Background] Miao H, Dong Y, Zhang Y, Zheng H, Shen Y, Crosby G, Culley DJ, Marcantonio ER, Xie Z. Anesthetic Isoflurane or Desflurane Plus Surgery Differently Affects Cognitive Function in Alzheimer's Disease Transgenic Mice. Mol Neurobiol. 2018 Jul;55(7):5623-5638. doi: 10.1007/s12035-017-0787-9. Epub 2017 Oct 6. PMID 28986748
- [Background] He J, Huang B, Zhang K, Liu M, Xu T. Long non-coding RNA in cervical cancer: From biology to therapeutic opportunity. Biomed Pharmacother. 2020 Jul;127:110209. doi: 10.1016/j.biopha.2020.110209. Epub 2020 May 20. PMID 32559848
- [Background] Lu G, Zhao W, Rao D, Zhang S, Zhou M, Xu S. Knockdown of long noncoding RNA WNT5A-AS restores the fate of neural stem cells exposed to sevoflurane via inhibiting WNT5A/Ryk-ROS signaling. Biomed Pharmacother. 2019 Oct;118:109334. doi: 10.1016/j.biopha.2019.109334. Epub 2019 Aug 16. PMID 31545269
- [Background] Zhao Y, Ai Y. Overexpression of lncRNA Gm15621 alleviates apoptosis and inflammation response resulting from sevoflurane treatment through inhibiting miR-133a/Sox4. J Cell Physiol. 2020 Feb;235(2):957-965. doi: 10.1002/jcp.29011. Epub 2019 Jul 2. PMID 31264218
- [Background] Niu X, Pu S, Ling C, Xu J, Wang J, Sun S, Yao Y, Zhang Z. lncRNA Oip5-as1 attenuates myocardial ischaemia/reperfusion injury by sponging miR-29a to activate the SIRT1/AMPK/PGC1alpha pathway. Cell Prolif. 2020 Jun;53(6):e12818. doi: 10.1111/cpr.12818. Epub 2020 May 28. PMID 32468629
- [Background] Tu Y, Zhu M, Wang Z, Wang K, Chen L, Liu W, Shi Q, Zhao Q, Sun Y, Wang X, Song E, Liu X. Melatonin inhibits Muller cell activation and pro-inflammatory cytokine production via upregulating the MEG3/miR-204/Sirt1 axis in experimental diabetic retinopathy. J Cell Physiol. 2020 Nov;235(11):8724-8735. doi: 10.1002/jcp.29716. Epub 2020 Apr 23. PMID 32324260
- [Background] Wang S, Han X, Mao Z, Xin Y, Maharjan S, Zhang B. MALAT1 lncRNA Induces Autophagy and Protects Brain Microvascular Endothelial Cells Against Oxygen-Glucose Deprivation by Binding to miR-200c-3p and Upregulating SIRT1 Expression. Neuroscience. 2019 Jan 15;397:116-126. doi: 10.1016/j.neuroscience.2018.11.024. Epub 2018 Nov 26. PMID 30496821
- [Background] Sun LY, Li XJ, Sun YM, Huang W, Fang K, Han C, Chen ZH, Luo XQ, Chen YQ, Wang WT. LncRNA ANRIL regulates AML development through modulating the glucose metabolism pathway of AdipoR1/AMPK/SIRT1. Mol Cancer. 2018 Aug 22;17(1):127. doi: 10.1186/s12943-018-0879-9. PMID 30134922
- [Derived] Jin D, Ma Y, Ji Y, Ge S. Impact of desflurane versus isoflurane on early cognitive function of the elderly undergoing lumbar surgery: a randomized clinical trial. BMC Anesthesiol. 2025 Dec 9;25(1):605. doi: 10.1186/s12871-025-03493-1. PMID 41366726